CLINICAL TRIAL: NCT01358305
Title: A Randomized, Controlled Double Blind Acute Study: Effects of Protein Blends on Muscle Protein Synthesis and Breakdown
Brief Title: Protein Blends (Soy, Whey and Casein) for Muscle Synthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DuPont Nutrition and Health (Industry)
Collaborators: University of Texas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: CRC-D-176
Record Dates: First submitted 2011-05-19; First posted 2011-05-23 (Estimated); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Muscle Synthesis
Keywords: muscle; synthesis; mTOR; antioxidant; inflammatory markers; soy protein; whey; casein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Whey Protein Isolate (Active Comparator)
  Interventions: Other: Protein Blend
- Protein Blend (soy, whey and casein) (Experimental)
  Interventions: Other: Protein Blend

INTERVENTIONS:
Other: Protein Blend — Single intake of approximately 20 grams of total protein

SUMMARY:
Soy protein is a high quality, plant-based protein that is comparable to milk, meat and eggs. Soy protein has a digestion rate (intermediate) compared to whey (fast) and casein (slow). This intermediate rate may allow soy protein to have an extended window of muscle protein synthesis that has not been monitored in previous studies. While most of the sports nutrition "recovery" products are dairy-based protein blends (high in branched-chain amino acids), soy protein offers additional benefits that can make an important contribution to these types of sports nutrition products. Soy protein contains approximately 300% more arginine and 30% more glutamine compared to whey protein and these two amino acids may bring additional benefits (immunity and hydration, respectively) to athletes. A "blend" of high-quality proteins (soy and dairy) may be the optimal sports nutrition product for athletes to consume following training.

ELIGIBILITY:
Inclusion:

1. Age 18-35 yrs
2. Stable body weight for at least 1 year

Exclusion criteria will be:

1. Exercise training (>2 weekly sessions of moderate to high intensity aerobic or resistance exercise)
2. Significant heart, liver, kidney, blood, or respiratory disease
3. Peripheral vascular disease
4. Diabetes mellitus or other untreated endocrine disease
5. Active cancer (all groups) and history of cancer (groups potentially randomizable to rapamycin)
6. Acute infectious disease or history of chronic infections (e.g. TB, hepatitis, HIV, herpes)
7. Recent (within 6 months) treatment with anabolic steroids, or corticosteroids.
8. Alcohol or drug abuse
9. Tobacco use (smoking or chewing)
10. Malnutrition (BMI < 20 kg/m2, hypoalbuminemia, and/or hypotransferrinemia)
11. Obesity (BMI > 30 kg/m2)
12. Low hemoglobin levels (below normal values)
13. Food allergies
14. Taking dietary supplements such as green tea, etc.
15. Currently on a high-soy diet (consuming >2 servings of soy per day)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2011-01; Primary Completion 2012-08 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Muscle Protein Synthesis or Fractional synthesis rate (FSR) | baseline, 3 hours, 5 hours
  The fractional synthesis rate (FSR) of mixed muscle proteins will be calculated from the incorporation rate of L-[ring-13C6]Phenylalanine into the mixed muscle proteins, and the free-tissue phenylalanine enrichment.

SECONDARY OUTCOMES:
oxidative and inflammatory markers | baseline, 3 hours, 5 hours
  Proteins will be assessed that are markers of oxidative damage and inflammation (NFkB, IL-1, IL-6) and proteolysis (MuRF, MAFBx).
Phosphorylation of protein in muscle protein signaling pathways | baseline, 3 hours, 5 hours
  Phosphorylation of mTOR, 4E-BP1, S6K1, S6, and eEF2 will be measured using Western blot techniques as previously described.

CONTACTS AND LOCATIONS:
Overall Officials: Ratna Mukherjea, PhD, Principal Investigator — Solae, LLC; Mark B Cope, PhD, Principal Investigator — Solae, LLC; Blake B Rasmussen, PhD, Principal Investigator — UTMB
Locations (1):
- UTMB General Clinical Research Center, located in the John Sealy Hospital, Galveston, Texas, United States

REFERENCES:
- [Derived] Reidy PT, Walker DK, Dickinson JM, Gundermann DM, Drummond MJ, Timmerman KL, Fry CS, Borack MS, Cope MB, Mukherjea R, Jennings K, Volpi E, Rasmussen BB. Protein blend ingestion following resistance exercise promotes human muscle protein synthesis. J Nutr. 2013 Apr;143(4):410-6. doi: 10.3945/jn.112.168021. Epub 2013 Jan 23. PMID 23343671